CLINICAL TRIAL: NCT05292222
Title: A Single Arm Study of Resting State Functional Magnetic Resonance Imaging (Rs-fMRI)-Guided Theta Burst Stimulation (TBS) in Early-Stage Alzheimer's Disease (AD)
Brief Title: Transmagnetic Stimulation Pilot in Early Stage Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A21-251
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Results first posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer Disease
Keywords: transmagnetic stimulation; functional MRI guided Theta Burst Stimulation; Early Stage
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Intermittent theta burst stimulation (Experimental): All subjects will receive treatment with intermittent theta burst stimulation (iTBS). There will be a total of 5 treatments over a 2-week period. All subjects will receive iTBS to the right TGd region. TBS treatment will also be provided for two additional sites within the large-scale brain networks (LSBNs) that is found to contain the greatest number of connectivity anomalies. Total participation will be 10-12 weeks.
  Interventions: Device: Intermittent theta burst stimulation

INTERVENTIONS:
Device: Intermittent theta burst stimulation — MagVenture TMS Therapy with theta burst stimulation. Resting motor threshold: 80%; Number of pulses per session: 1200 pulses; Inter-train interval: 8 seconds; Pulse frequency in burst: 50 Hertz
  Other Names: Transmagnetic stimulation; MagVenture

SUMMARY:
Alzheimer's disease (AD) is a progressive neurodegenerative condition affecting 6.2 million individuals in the United States, resulting in an annual cost of care of $305 billion. AD is functionally characterized by progressive degeneration of large-scale brain networks (LSBNs), including the default mode network (DMN) presumably from the deposition of amyloid plaques and neurofibrillary tangles. Available FDA-approved medications for AD such as donepezil and memantine offer limited benefit and modest impact on quality of life. In combination with resting state functional MRI (rs-fMRI), transcranial magnetic stimulation (TMS) with intermittent theta burst stimulation (iTBS) offers a non-invasive alternative to pharmacotherapy in persons with AD. We propose a pilot trial using rs-fMRI to target dysfunctional LSBNs in early stage AD.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of Mild Cognitive Impairment (MCI)/mild AD
* Evidence for Central Nervous System (CNS) amyloidosis (e.g., Amyloid positron emission tomography (PET) or cerebrospinal fluid (CSF) biomarkers consistent with AD)
* Prior brain imaging performed
* Mini-Mental State Examination (MMSE) >24
* Clinical Dementia Rating (CDR) Scale 0.5-1
* Stable dose of cholinesterase inhibitors and memantine for at least one month
* Subjects are between 40-90 years of age

Exclusion Criteria:

* Non-AD dementia including, but not limited to, Lewy body dementia, frontotemporal dementia, vascular dementia, Jakob-Creutzfeldt disease, etc.
* Inability to tolerate rs-fMRI
* Contraindication of rs-fMRI due to implants or metal
* Seizure disorder

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhavani Kashyap, MBBS, PhD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
No identifiable data will be shared with other researchers.

REFERENCES:
- [Derived] Kashyap B, Hanson LR, Gustafson SK, Barclay T, Howe CM, Sherman SJ, Hungs M, Rosenbloom MH. Open label pilot of personalized, neuroimaging-guided theta burst stimulation in early-stage Alzheimer's disease. Front Neurosci. 2024 Dec 9;18:1492428. doi: 10.3389/fnins.2024.1492428. eCollection 2024. PMID 39717698

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 participants screen failed with a low MMSE, 1 participant withdrew before receiving any treatment.
Period: Overall Study
Arm/Group | Intermittent Theta Burst Stimulation
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intermittent Theta Burst Stimulation
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Mini Mental Status Examination (MMSE) [Mean (Standard Deviation); unit: units on a scale] — The MMSE measures cognitive and mental status. Total score. Range [0-30]. Lower score is indicative of more cognitive impairment.
  units on a scale | 26.3 (1.2)
Clinical Dementia Rating (CDR) Scale [Mean (Standard Deviation); unit: units on a scale] — The global CDR is a scale used to quantify the severity of dementia symptoms. Range [0-3]. A higher score is indicative of more severe dementia symptoms.
  units on a scale | 0.5 (0)
Education Level [Count of Participants; unit: Participants]
  Bachelors/Associates | 6
  Masters/PhD | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Connectivity Measure of the TGd Parcellations.
Description: Assessed by calculating the difference and standard deviation between follow-up and baseline of number of abnormal connections of the TGd parcellation. Range: 0-378. There are 378 possible connections of the parcellation. Higher values indicate more abnormal connections of the TGd parcellation pre and post-treatment. The change in the number of abnormal connections of the parcellation is reported.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: abnormal connections
Arm/Group | Intermittent Theta Burst Stimulation
Number analyzed (Participants) | 10
abnormal connections | 0.5 (25)

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | Intermittent Theta Burst Stimulation
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intermittent Theta Burst Stimulation (N=10)
Facial or jaw twitching at RTGd site (Musculoskeletal and connective tissue disorders) | 10
Headache (General disorders) | 1
tearing of the eye (Eye disorders) | 1
facial twitching at other sites (Musculoskeletal and connective tissue disorders) | 2
Scalp pain (Musculoskeletal and connective tissue disorders) | 1
Altered consciousness (General disorders) | 1 — Happened between treatment days. Participant completed the treatment following evaluation for seizure and cardiac conditions with negative findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT05292222/Prot_SAP_000.pdf